CLINICAL TRIAL: NCT06207461
Title: Effects of Traditional Chinese Acupoint Massage on Gastrointestinal Function Recovery of ICU Patients: a Single-center, Prospective, Non-blind, Randomized Study
Brief Title: Traditional Chinese Acupoint Massage for Gastrointestinal Function Recovery
Status: Withdrawn | Type: Observational
Why Stopped: Medical ethics have yet to be passed
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jiancheng Zhang, Prof. Jiancheng Zhang, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: ZJC202401
Record Dates: First submitted 2023-12-03; First posted 2024-01-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Traditional Chinese Acupoint Message; Intestinal Barrier; Gastrointestinal Dysfunction
Keywords: Acupoint massage; Gastrointestinal dysfunction; Gastrointestinal function recovery; Intensive care unit; Intestinal barrier

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- massage group: patients with gastrointestinal function injury caused by medical diseases or with high risk of malnutrition who got massage
- non-massage group: patients with gastrointestinal function injury caused by medical diseases or with high risk of malnutrition who got no massage

SUMMARY:
Patients in the intensive care unit (ICU) are often at risk of gastrointestinal dysfunction and malnutrition. Gastrointestinal dysfunction was associated with poor clinical outcomes, including prolonged mechanical ventilation, prolonged ICU stay and increased 90-day mortality.

There have been some clinical studies investigating the effects of traditional Chinese acupoint massage, acupuncture, or moxibustion of 7 acupoints (Zhongwan Point (CV12), Tianshu Point (ST25), Qihai Point (CV6), Zusanli point (ST36), Shangjuxu Point (ST37), Neiguan Point (PC6) and Hegu Point (LI4)) on gastrointestinal function recovery. Gastrointestinal dysfunction could be improved by stimulating single acupoint or combining multiple acupoints, and the effects of combined stimulation of multiple acupoints was better for the improvement of gastrointestinal dysfunction.

This project aims to study the effects of traditional Chinese acupoint massage, acupuncture, or moxibustion of 7 acupoints (Zhongwan Point (CV12), Tianshu Point (ST25), Qihai Point (CV6), Zusanli point (ST36), Shangjuxu Point (ST37), Neiguan Point (PC6) and Hegu Point (LI4)) on the 28-day survival, and the gastrointestinal function recovery in critically ill patients with with gastrointestinal dysfunction caused by medical diseases and critically ill patients with high risk of malnutrition in ICU, and to observe their effects on the recovery of gastrointestinal barrier function by measuring the serum intestinal fatty acid binding protein (iFABP), citrulline, diamine oxidase (DAO) and D-lactic acid. Studies have shown that serum iFABP, citrulline, DAO and D-lactic acid could reflect the intestinal barrier function of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-80 years old without restriction of gender, race, religion, creed or nationality;
2. Patients with high risk of malnutrition due to gastrointestinal dysfunction caused by medical diseases, and AGI score Ⅰ-Ⅱ or NRS 2002 score ≥3 points;
3. Patients with hospital stay longer than 120 hours;
4. Willing to participate in this trial.

Exclusion Criteria:

1. Patients with abdominal open trauma;
2. Defects, infections or lesions in the skin near the acupoints；
3. Patients with abdominal tumor or large amount of abdominal fluid;
4. Patients with AGI score Ⅲ or above;
5. Pregnant patients;
6. Patients with Child-Pugh grade B and grade C liver function
7. Unable or unwilling to provide informed consent or poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients at high risk of malnutrition due to gastrointestinal functional impairment caused by medical diseases in the ICU, and AGI grade I-II or NRS 2002 score ≥3.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
28-day survival rate (%) | Up to 4 weeks
  Survival at 28 days after hospitalization
Ultrasound assessment of gastrointestinal function: ACF (times/min) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Antral contraction frequency (ACF): In semi-recumbent position at 45°, infuse the stomach with 300ml of warm water. Within 6 minutes after infusion, divide the number of antral contractions by 3.
Ultrasound assessment of gastrointestinal function: ACA (%) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Antral contraction amplitude (ACA): Measure the area during 3 maximum relaxations (S relaxation) and minimum contractions (S contraction), calculate the change in antral area (ΔS = S relaxation - S contraction), and take the average of 3 measurements. Antral contraction amplitude: ΔS/S relaxation.
Ultrasound assessment of gastrointestinal function: MI | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Motility index (MI): ACF × ACA.
Ultrasound assessment of gastrointestinal function: GET (min) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Gastric emptying time (GET): In semi-recumbent position at 45°, infuse the stomach with 300ml of warm water. Use the maximum antral relaxation as the standard and measure the area every 5 minutes until the liquid in the antrum is emptied. The time it takes for the gastric antrum to empty is GET.
Ultrasound assessment of gastrointestinal function: intestinal wall thickness (mm) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Intestinal wall thickness of Jejunum/Ileum/Colon: Refers to the distance between the serosal and mucosal surfaces of the intestinal wall. The normal thickness of the small intestine is 2-3mm, and >3mm may indicate thickening of the intestinal wall; the thickness of the colon wall is approximately 3-4mm, and >5mm may suggest thickening of the intestinal wall. Attention should be paid to the colon pocket and the plica structure on the colon wall.
Ultrasound assessment of gastrointestinal function: intestinal diameter (cm) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Intestinal diameter of Jejunum/Ileum/Colon: When not under pressure, the measurement of the width of the small intestine often refers to the distance between the mucosal surfaces of the intestinal wall. The intestinal lumen width of the small intestine (jejunum/ileum) is generally <2cm, and >3cm may indicate intestinal dilation; the internal diameter of the colon is generally <5cm.
Ultrasound assessment of gastrointestinal function: intestinal motility | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Intestinal motility of Jejunum/Ileum/Colon (yes or no): Under normal circumstances, intestinal movement can be clearly judged at the ultrasound interface. When the intestine is filled with gas or accompanied by intestinal dilation, intestinal motility can be judged by the "creeping gas sign" of the gas or the movement of the contents. In addition, attention should be paid to the intestinal motility caused by the pressure on the intestinal tube when moving the probe.

SECONDARY OUTCOMES:
Daily amount of enteral nutrition feeding (ml) | Within 5 days after study inclusion
  Daily amount of enteral nutrition feeding
Daily gastric residual volume (ml) | Within 5 days after study inclusion
  Daily gastric residual volume
Serum levels of intestinal fatty acid binding protein (iFABP, ng/ml) | 0, 72 and 120 hours after study inclusion
  Serum levels of iFABP measured by ELISA.
Serum levels of citrulline (μmol/L) | 0, 72 and 120 hours after study inclusion
  Serum levels of citrulline measured by ELISA.
Serum levels of diamine oxidase (DAO, U/L) | 0, 72 and 120 hours after study inclusion
  Serum levels of DAO measured by ELISA.
Serum levels of D-lactic acid (mmol/L) | 0, 72 and 120 hours after study inclusion
  Serum levels of D-lactic acid measured by ELISA.
Superior mesenteric artery resistance index | 0, 72 and 120 hours after study inclusion
  Superior mesenteric artery resistance index evaluated by ultrasound
Intra-abdominal pressure (IAP) (mmHg) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Intra-abdominal pressure (IAP)
Diarrhea | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Yes (numbers) or No
Alimentary tract hemorrhage | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Yes (numbers) or No
Prealbumin concentration (g/L) | 0, 72 and 120 hours after study inclusion
  Serum levels of prealbumin
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
ICU length of stay (days) | Up to 4 weeks
  ICU length of stay
In-hospital mortality (%) | Up to 4 weeks
  Mortality rate during hospitalization
Peripheral venous blood CRP concentration (mg/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  CRP level measured by blood routine examination
Peripheral venous blood hemoglobin concentration (g/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Hemoglobin level measured by blood routine examination
Absolute number of white blood cells in the peripheral venous blood (number/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Absolute number of white blood cells measured by blood routine examination
Absolute number of platelets in the peripheral venous blood (number/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Absolute number of platelets measured by blood routine examination
Absolute number of lymphocytes in the peripheral venous blood (number/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Absolute number of lymphocytes measured by blood routine examination
Whole blood pH | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Arterial pH measured by blood gas analysis
Arterial PaO2 (mmHg) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Arterial PaO2 measured by blood gas analysis
Arterial PaCO2 (mmHg) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Arterial PaCO2 measured by blood gas analysis
Arterial bicarbonate (mmol/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Arterial bicarbonate measured by blood gas analysis
Arterial lactic acid (mmol/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Arterial lactic acid measured by blood gas analysis
Peripheral venous blood albumin concentration (g/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Albumin level measured by Blood biochemical examination
Peripheral venous blood total bilirubin concentration (μmol/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Total bilirubin level measured by Blood biochemical examination
Peripheral venous blood bound bilirubin concentration (μmol/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Bound bilirubin level measured by Blood biochemical examination
Peripheral venous blood creatinine concentration (μmol/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  Creatinine level measured by Blood biochemical examination
Peripheral venous blood ALT concentration (U/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  ALT level measured by Blood biochemical examination
Peripheral venous blood AST concentration (U/L) | 0, 24, 48, 72, 96 and 120 hours after study inclusion
  AST level measured by Blood biochemical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China